CLINICAL TRIAL: NCT02947243
Title: Decreasing REcurrent Pain and Anxiety in Medical Procedures With a Pediatric Population: Trial
Acronym: DREAM-T
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Major changes to protocol (new study design and comparator)
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1383
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Pain; Burns; Child; Anxiety
Keywords: Virtual reality; Immersive distraction; Oculus rift; Virtual world; Virtual environment; Procedural pain; Procedural anxiety; Acute pain; Pain management; Anxiety; Children, Child; Kid, Kids; Pediatric, Pediatrics; Young children; Burns; Burn injuries; Burn unit; Physiotherapy; Physical therapy; Burn dressing; Dressing change; Non-pharmacological, nonpharmacological; Clinical Research; Nursing Practice
MeSH Terms: conditions — Pain; Burns; Anxiety Disorders; Pain, Procedural; Acute Pain; Agnosia; Deafness, Autosomal Recessive 1A | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pharmacological treatment (Active Comparator): Standard pharmacological treatment (including Morphine) according to the unit's protocol and adjusted to each participant's age, weight and condition by the anesthetist and pain clinic nurse.
  Interventions: Drug: Morphine
- VR distraction via Oculus Rift (Experimental): In addition to standard pharmacological treatment, Virtual reality distraction through the use of Oculus Rift® will be used as the experimental intervention.
  Interventions: Device: VR distraction via Oculus Rift

INTERVENTIONS:
Device: VR distraction via Oculus Rift — In addition to standard pharmacological treatment, Virtual reality distraction through the use of Oculus Rift® will be used as the experimental intervention. The Oculus Rift (Consumer version) is made of two Oled panels with a resolution of 1200p running at 90Hz. It has very effective 360 degree positional tracking and integrated 3D audio. These combine to produce a high level of immersion, with high photorealism while maintaining the low latency necessary to induce presence and prevent cybersickness. The child, depending on the burn site, will have the opportunity to interact with the game. Video games, approved by healthcare professionals with extensive experience in pediatrics, will be adapted for children and tailored to minimize cyber sickness.
  Arms: VR distraction via Oculus Rift
Drug: Morphine — As per unit's protocol
  Other Names: Standard pharmacological treatment
  Arms: Standard pharmacological treatment

SUMMARY:
Children with burn injuries experience severe pain intensity during medical procedures despite the increasing doses of analgesics. Current guidelines on pediatric procedural pain management recommend the combination of non-pharmacological and pharmacological interventions to enhance pain management and decrease the numerous side effects of analgesics. Virtual reality (VR) has gained growing consideration as a non-pharmacological method as it engages multiple senses and allows interactions with a virtual world. Oculus Rift ® is a new technology in VR that provides more immersiveness, at a relatively low cost, and could probably improve the management of pain and anxiety in burn care. It also has the potential, with appropriate custom software designed for burn pediatric patients, to reduce the cybersickness symptoms (nausea, dizziness) associated with VR. To the knowledge of the investigators, none of the pediatric hospitals across Canada have tested VR as a method of pain and anxiety management in children with burn injuries. Overall hypotheses: VR distraction via Oculus Rift ® could be an effective method to relieve pain, and anxiety, as well as a less traumatizing hospital experience, while promoting a more humanistic care environment by combining new technologies (VR via Oculus Rift ®) to standard analgesic interventions administered to these children. The expected results will have a direct effect on physical (pain) and psychological (anxiety, pain memories) health of the child. In addition, clinical implications may include other indicators of quality of care and economic benefits such as a wider range of motion of burned limbs and reduction in dosage of opioids and anxiolytic drugs administered.

DETAILED DESCRIPTION:
1. BACKGROUND:

   Burn injuries are the leading cause of morbidity and mortality in children. They are associated with a lot of pain that is difficult to treat and can impede recovery, cause high levels of anxiety and alter future pain behaviors, resulting at times in chronic pain, paresthesia, or depression. Pain can also decrease participation in treatments such as physiotherapy resulting in poor health outcomes. Beyond the immediate pain experience, children may develop memories that are accurate, positively or negatively estimated (i.e., remembering more or less pain, respectively, as compared to initial pain reports). The way that children's memories are framed is important for future pain coping and distress at subsequent painful experiences. Moreover, it has been shown that pharmacological and non-pharmacological pain management strategies may buffer children from developing such biases in pain memories. Procedural pain is still largely managed pharmacologically mostly through the use of opioids, benzodiazepines and other pharmacological agents which cause a lot of side effects and do not always provide sufficient pain reduction. In recent years, the effectiveness of multimodal approaches combining medication with non-pharmacological interventions for procedural pain relief has been highlighted. Distraction techniques engaging multiple senses may grab the child's attention more than the techniques that only engage one sense (e.g, music), hence, the increasing interest in more immersive and interactive methods of distraction such as VR.

   VR is an active distraction method that allows the user to interact with an immersive environment generated by a computer stimulating different senses. A review of studies on VR, mostly conducted with adult burn patients, showed a 35 to 50% reduction in procedural pain while using VR. However, despite promising results, the use of VR in healthcare settings has been limited, mainly due to its high cost. Reviews have highlighted the need for more research but mostly for the development of more portable, less expensive and more developed VR systems that would promote pain reduction during burn procedures especially for children with burn injuries who are considered one of the most challenging burn populations. However, there has been a breakthrough in technology since 2014 when big scale companies started investing in VR development for commercial gaming. Facebook purchased the Oculus Rift® for mass production allowing access to the latest technology in VR at a relatively low cost. Oculus Rift® is a VR tool that provides a wide field of view, high resolution display, integrated 3D audio and motion detection. In addition, its highly immersive properties could help achieve more analgesia compared to other VR techniques as a review has shown that the sense of presence influences the effectiveness of VR-based analgesia. The sense of presence is a subjective psychological state of consciousness of being in the virtual world whereas immersiveness refers to the physical environment that could be quantified by measuring the field of view or the peripheral vision in the VR goggles. The availability of inexpensive yet highly immersive VR googles such as Oculus Rift® could increase the use of VR in pain management and burn settings while significantly improving its cost effectiveness. A single case study assessed the feasibility of a VR intervention via Oculus Rift® in one child of 11 years old with burn injuries during occupational therapy. The study showed a reduction in pain intensity and pain unpleasantness experienced by the patient, without any side effects. To the knowledge of the investigators, no other studies have tested the distraction via Oculus Rift® for procedural pain management in children with burn injuries undergoing painful physiotherapy treatments.
2. AIM:

   The aim of this study is to assess the effect of distraction by VR via Oculus Rift® for the relief of procedural pain, anxiety and decrease memory of pain in children with burn injuries.

   Primary Research Question: In children aged 7 to 18 years, who have suffered burn injuries, does VR distraction via Oculus Rift® combined with analgesics provide better pain relief during painful procedures including dressing changes and physiotherapy than standard pharmacological treatment alone?

   Secondary Research Questions: a) In children aged 7 to 18 years, who have suffered burn injuries, does VR distraction via Oculus Rift® combined with analgesics provide better anxiety relief during dressing change and physiotherapy than standard pharmacological treatment alone? b) Does the use of VR distraction lead to less distressing memories of pain than standard pharmacological treatment alone? c) Does the use of VR distraction reduce the dose and side effects of analgesics used during burn wound dressing changes and physiotherapy in children?
3. HYPOTHESES

   1. VR distraction via Oculus Rift® combined with analgesics is more effective than standard treatment (analgesics alone) to manage procedural pain of children with burn injuries.
   2. VR distraction via Oculus Rift® combined with analgesics is more effective than standard treatment (analgesics alone) on procedural anxiety of children with burn injuries.
   3. VR distraction via Oculus Rift® combined with analgesics will lead to less distressing memories of pain than standard treatment (analgesics alone) in children with burn injuries
4. METHODS 4.1 Design. One-group within subject/crossover study design. Given the difficulty of ensuring a single or a double-blind condition, and in order to limit the interpersonal variability between participants, each child will serve as their own control and will receive both standard and experimental treatments during the same treatment session through a randomized order.

4.2 Sample and Setting. Participants will be recruited through convenience sampling upon admission to the surgical-trauma burn unit at CHU Ste-Justine, Montreal (Qc), Canada. For a statistical power of 80%, an alpha of 0.05, and a significant difference of two points on a 0 to 10 on the NRS pain scale, the size of the total desired sample is 40 participants who will serve as their own controls. The setting of the study is the main referral center for pediatric burns in Quebec. It receives nearly 60 admissions during the time of the year when there is a higher incidence of burns (April to October) and over all close to 100 admissions per year. One third of the total admissions are aged 7 years and older. Given a possible census of 33 admissions per year, it appears feasible to recruit around 40 patients over a period of two years. This is also the reason behind the choice of the design which would be the most feasible given the total population available for recruitment.

.3 Interventions. A) Standard pharmacological treatment B) Standard treatment in addition to Virtual Reality distraction via Oculus Rift

4.4. Measures. Pain, anxiety and comfort measures will be taken before the treatment (physiotherapy or dressing change) session (T1) (for expectancy and baseline state), after the first sequence of the session (T2) and after the second sequence of the session (T3). Healthcare professionals will be asked to fill an anonymous satisfaction questionnaire 30 minutes after the end of the session (T4). Memories of pain/anxiety will be assessed at least 24 hours after each procedure (T5).

4.5 Study proceedings. Physiotherapy and dressing change sessions typically last between 10 and 20 minutes. The duration will be divided in two sequences of the same duration (5 to 10 minutes) where the participant receives the same treatment (range-of-motion exercises for physiotherapy or wound cleaning and gauzes application for dressing changes) by the same healthcare professional (physiotherapist or nurse). For one sequence, only the standard pharmacological treatment will be administered and for the other sequence, patients will receive the standard pharmacological treatment in addition to the virtual reality distraction via OR. The order of sequences will be randomized.

4.6 Data analysis plan. Multivariate Analyses and quantitative comparisons will be conducted within and between subjects for the dependent variables for repeated measures. The mean difference in pain scores of patients at each time-period will be compared using a paired t-test. Since the use of rescue medication is a potential indication of a treatment failure, the primary analysis will be supplemented by an analysis comparing the proportion of patients receiving rescue medication anytime during the procedure. Interpretation of the primary analyses will be made with reference to the data regarding rescue medication use. Data collected on dichotomous variables will be analyzed using a chi-square test and post-hoc analyses if the results are statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* suffer from a burn injury requiring wound dressing change or physiotherapy
* presence of a consenting parent who can understand, read and write either French or English

Exclusion Criteria:

* requiring intensive care
* having a diagnosed cognitive impairment
* are unconscious or intubated during dressing change or physiotherapy
* suffer from epilepsy (considering the nature of the intervention)
* allergic to opioids or other analgesics used for standard pharmacological treatment
* having burn injuries on the face preventing the use of the Oculus Rift headset

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mean Pain Score | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Numerical Rating Scale (NRS) ranging from 0 to 10; 0=no pain to 10=pain as bad as it could be

SECONDARY OUTCOMES:
Pain Experience | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Graphic Rating Scale (GRS) consisting of seven items to measure the cognitive, the affective and the sensory components of pain
Expected Anxiety | Baseline (T1)
  Children's Fear Scale (CFS)
Experienced Anxiety | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Children's Fear Scale (CFS)
Satisfaction Level | T4: 30 minutes after the procedure
  Satisfaction questionnaire developed by the team
Side Effects | T4: 30 minutes after the procedure
  Nausea, vertigo or other side effects related to the use of Oculus Rift
Comfort Level | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Behavioural observation scale of comfort level for child burn victims (OCCEB-BECCO)
Pain Memory | 24 hours after the procedure (T5)
  A measure of the child's memory of pain using the same measure (NRS) administered during the initial data collection to assess this construct
Anxiety Memory | 24 hours after the procedure (T5)
  A measure of the child's memory of anxiety using the same measure (CFS) administered during the initial data collection to assess this construct
Range Of Motion | Baseline (T1); T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  (only for physiotherapy sessions) Using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste. Justine, Montreal, Quebec, Canada